CLINICAL TRIAL: NCT06289803
Title: The Application of Probe Confocal Laser Endomicroscopy in Pancreatic Tumor Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Huadong Hospital of FudanU
Record Dates: First submitted 2023-10-17; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer; Diagnosis; Pancreatoduodenectomy; Distal Pancreatectomy
Keywords: pancreatic cancer; confocal laser endomicroscopy; resection margin; diagnosis; radical resection
MeSH Terms: conditions — Pancreatic Neoplasms; Disease; Margins of Excision

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with pancreatic tumours will undergo surgical resection, and PCLE will be used for identifying the behaviour of tumours (benign or malignant neoplasms) and predicting the status of resection margin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients who accept the scan of pCLE (Experimental)
  Interventions: Device: probe confocal laser endomicroscopy

INTERVENTIONS:
Device: probe confocal laser endomicroscopy — probe confocal laser endomicroscopy will be used to identify the tumor behavior

SUMMARY:
Aim of the study: To evaluate the value of Probe Confocal Laser Endomicroscopy (PCLE) in surgery for pancreatic tumor.

Methods:

Patients who are diagnosed with pancreatic tumor based on preoperative radiographic findings and will undergo radical resection are included in this clinical study. PCLE will be used in surgery to identify tumor is malignant or not, and surgeons will decide procedures of surgery based on outcomes of PCLE. In this present study, clinical trials will be divided into two phases. In the first phase, based on the definitive postoperative pathologic diagnosis, characteristic imaging structures that were collected by PCLE will be identified and primary diagnostic imaging criteria for pancreatic cancer would be developed. In the second phase, this criterion will be used for rapid intraoperative diagnosis of pancreatic cancer and predicting status of resection margin. In addition, accuracy of PCLE will be verified based on postoperative pathologic reports.

DETAILED DESCRIPTION:
Accurately identifying benign and malignant pancreatic tumor is a challenge for surgeons. Although pathological reports are the golden standard for determining the behaviour of pancreatic tumor, it's too late for patients with benign tumor because excessive resection has been performed. Unnecessary resection will cause great harm for those patients. Freezing microtomy during surgery is a method to distinguish the essence of the tumor in surgery, but it's still time-consuming and inaccurate. Recently, lots of studies reported that Probe Confocal Laser Endomicroscopy (PCLE) is potentially effective tool for determining the nature of pancreatic tumor with high sensitivity and specificity. However, there are no imaging criteria regarding PCLE for the diagnosis of pancreatic cancer, and it's underused in intraoperative scenes of pancreatic surgery for quickly recognizing malignant pancreatic tumor. The aim of the present study is to summarize the special structures of image collecting by PCLE and evaluate its practical value. If PLCE is proven to be as diagnostic efficiency as pathology in this study, patients who diagnosed with pancreatic benign tumor by PCLE will opt for local excision rather than pancreaticoduodenectomy or distal pancreatectomy. What's more, if patients are diagnosed with pancreatic cancer by PCLE, example pancreatic adenocarcinoma, they will undergo radical resection (the Whipple procedure or distal pancreatectomy). In addition, PCLE will be used for predicted the status of resection margin. If positive margin status are detected by scanning the wound of tumor, surgeons will expand the resection.

ELIGIBILITY:
Inclusion Criteria:

1. patients are diagnosed with pancreatic neoplasms based on preoperative radiographic findings and auxiliary examination results, and they will undergo pancreatoduodenectomy or distal pancreatectomy.
2. Patients who have no serious abnormalities of blood system, heart and lung function and immune deficiency and can tolerate surgery.
3. Patients who are not allergic to fluorescein sodium will be included.

Exclusion Criteria:

1. Patients accompanied by other systemic malignancies.
2. Central nervous system disease, mental disease, unstable angina pectoris, congestive heart failure, serious arrhythmia and other uncontrollable serious diseases, unable to tolerate surgery.
3. Patients who have had definitive pathologic diagnosis before surgery will be excluded.
4. Any condition that may impair the safety of patients or the integrity of research data, including serious medical risk factors, medical conditions, and laboratory abnormalities.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic efficacy | up to 30 postoperative days
  Sensitivity(Se), Specificity(Sp), Accuracy, positive predictive value (PPV), Negative predictive value (NPV),

SECONDARY OUTCOMES:
Rate of R0 resection | up to 30 postoperative days
  Percentage of R0 margins in pancreatic cancer surgery by using PCLE

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China